CLINICAL TRIAL: NCT04172337
Title: A Randomized Controlled Trial Testing the Effects of Singapore's Front-of-Pack Healthier Choice Symbol Label With or Without a Physical Activity Equivalent Label on Food Purchases and Measures of Diet Quality
Brief Title: Testing the Effects of Singapore's Front-of-Pack Healthier Choice Symbol Label With or Without a Physical Activity Equivalent Label
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Principal Investigator, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NMRC-HSRG-0060-2016
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Diabetes; Diet, Healthy
Keywords: nutrition; front-of-pack label; calories; online grocery store; Singapore; physical activity equivalent
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This will be a crossover study design with all participants exposed once to 3 shopping conditions (1xControl, 1x Arm 2 and 1x Arm 3) in random order. The total study duration for each participant is 3 weeks, with each participant spending 1 week in each shopping condition.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Using a within-person crossover design, participants were randomly assigned to one of six intervention sequences, which included the order of the three shops and when the actual purchase would take place, via random permuted blocks of size three with equal allocation for the six sequences (see Appendix Table A1) by a computer program. Participants were blinded to intervention allocation, which was allocated via the NUSMart system. Allocation results were recorded within NUSMart and all investigators, including the data analyst, were blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No labeling Control (No Intervention): Arm 1 was the Control condition, which did not display FOP labels on any products.
- HCS-only (Experimental): Arm 2 (termed HCS-only) displayed the HCS on eligible products, crossed referenced via the Health Promotion Board's HCS database (https://www.hpb.gov.sg/food-beverage/healthier-choice-symbol). Out of the 4,177 products available on NUSMart, 311 (7·45%) carried the HCS. This was comprised of 150 foods and 161 beverages.
  Interventions: Behavioral: Healthier Choice Symbol
- HCS+PAE (Experimental): Arm 3 displayed the HCS on eligible products as in Arm 2 and the PAE label on all products (termed HCS+PAE). PAE was calculated as the minutes required to burn off the calories of a single serving for a 73 kg person jogging at 8 km per hour.
  Interventions: Behavioral: Healthier Choice Symbol; Behavioral: Physical Activity Equivalent label

INTERVENTIONS:
Behavioral: Healthier Choice Symbol — The HCS is intended to improve diet quality by signaling to consumers which products are healthier options within a specific category (e.g., which are the healthier biscuits or the healthier beverages). Manufacturers must meet category-specific criteria before a product can display the HCS and an associated tagline. The labels were displayed at the bottom of the product images.
  Arms: HCS+PAE; HCS-only
Behavioral: Physical Activity Equivalent label — For the study, we designed a simple PAE logo (Appendix Figure A1) and added a description encoded into the NUSMart user interface to ensure that participants would understand the contents of the label. Participants saw the following description whenever their cursor hovered over the PAE label: "The Physical Activity Equivalent (PAE) refers to the number of minutes that a typical adult would need to jog to burn off the calories associated with one serving of the product." Previous studies have shown this labelling approach to be effective.
  The labels were displayed at the bottom of the product images.
  Arms: HCS+PAE

SUMMARY:
Poor diets are known risk factors for chronic diseases, and in recent years, food labelling has been increasingly sought-after as a cost-effective intervention to help stem the rising trend in chronic diseases.

In efforts to promote a healthy diet, the Singapore Health Promotion Board (HPB) supplements traditional nutrition labelling with the Healthier Choice Symbol (HCS), which identifies food items within a specific category of foods as healthier choices. The original logos were enhanced to include additional information focusing on particular macronutrients, taking one of two themes; it either indicates that a product contains more of a healthier ingredient, or less of a less healthy ingredient.

However, to date, no published studies have assessed the role of the original and enhanced HCS logos in influencing food choices. There is a lack of scientific evidence on the role of the existing symbols in assisting consumers make healthier food purchasing decisions. There are also concerns over the unintended consequences of health claims made based on a single aspect of nutrient content, without considering other aspects. That is the goal of this effort. Specifically, the investigators

propose to conduct the following:

Use a three arm randomized controlled trial (RCT) and an experimental fully functional web-based grocery store to assess the causal effect of the new HCS logos on measures of diet quality either alone, or in combination with a complementary front-of-package (FOP) label: Physical Activity Equivalents (PAEs), which provides information on how long one would need to engage in a certain activity (e.g., jogging) to burn off one serving of the product.

The investigators hypothesize that the greatest reduction in calories per serving (primary outcome) will occur in the HCS plus PAEs arm, followed by HCS only, and no logo control arm.

ELIGIBILITY:
Inclusion Criteria:

* Singapore residents
* 21 years of age and above
* Primary grocery shopper for the household

Exclusion Criteria:

* Not residing in Singapore
* Under 21 years of age
* Not the primary grocery shopper for the household

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in average calories per serving purchased per shopping trip | Once a week for three weeks
  Calories per serving (kCal per serving) is calculated by dividing the total number of calories purchased in the shopping trip by the total number of servings purchased. The average calories per serving purchased (kcal per serving) is based on mean standardized serving sizes within each subcategory.

SECONDARY OUTCOMES:
Proportion of HCS labelled products purchased (or would have been if not in control arm) per shopping trip | Once a week for three weeks
  Calories per Shopping Trip will be calculated as the sum of all purchased products' total calories.
Total Calories per shopping trip | Once a week for three weeks
  Total calories purchased in kcal.
Diet quality per shopping trip as measured by the Grocery Purchase Quality Index-2016 | Once a week for three weeks
  Diet quality per shopping trip as measured by the Grocery Purchase Quality Index-2016 (GPQI-2016). The Grocery Purchase Quality Index-2016 (GPQI-2016) contains 11 different food components with eight components scored based on adequacy and three moderation components. We followed the standard GPQI-2016 scoring methods by mapping NUSMart's subcategories to USDA food plan categories and then to the GPQI components. Each component was scored based on the deviation of the observed expenditure share of each component and the expected expenditure share, and the scores were totaled up to generate the final GPQI-2016 score (minimum possible score = 0, maximum possible score = 75) for each participant's weekly grocery order. A higher score indicates better diet quality of the grocery basket.
Diet quality per shopping trip as measured by weighted average Nutri-Score | Once a week for three weeks
  We applied the standard Nutri-Score algorithm to assign a grade to each product. This algorithm assigns a score of A to E based on nutritional quality, which we recoded to 5 to 1 and then calculated an average score for each participant's weekly grocery order (minimum possible score = 0, maximum possible score = 5), weighted by the number of servings of each product. A higher score indicates better diet quality of the grocery basket.
Sugar per serving per shopping trip | Once a week for three weeks
  Amount of sugar (g) per serving purchased based on mean standardized serving sizes within each subcategory.
Sodium per serving per shopping trip | Once a week for three weeks
  Amount of sodium (mg) per serving purchased based on mean standardized serving sizes within each subcategory.
Saturated fat per serving per shopping trip | Once a week for three weeks
  Amount of saturated fat (g) per serving purchased based on mean standardized serving sizes within each subcategory.
Calories per dollar spent per shopping trip | Once a week for three weeks
  Number of calories per dollar (kcal per dollar) spent

CONTACTS AND LOCATIONS:
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
We will make de-identified data used in the manuscript available to editors upon request either before or after publication for checking.
Supporting Information: Study Protocol, ICF
Time Frame: 10 years after study completion
Access Criteria: Reasonable request

REFERENCES:
- [Derived] Finkelstein EA, Doble B, Ang FJL, Wong WHM, van Dam RM. A randomized controlled trial testing the effects of a positive front-of-pack label with or without a physical activity equivalent label on food purchases. Appetite. 2021 Mar 1;158:104997. doi: 10.1016/j.appet.2020.104997. Epub 2020 Oct 13. PMID 33065191